CLINICAL TRIAL: NCT00905424
Title: A Phase 2, Multicenter, Randomized, Double-blind, Parallel-group, Placebo Controlled Exploratory Efficacy and Safety Study of SPD489 in Adults 18-55 Years With Major Depressive Disorder (MDD) as Augmentation Therapy to an Antidepressant
Brief Title: Exploratory Study of SPD489 in Adults With Major Depressive Disorder (MDD) as Augmentation Therapy to an Antidepressant
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Shire (Industry)
Responsible Party: Sponsor
Organization: Takeda (Industry)
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: SPD489-203
Record Dates: First submitted 2009-05-18; First posted 2009-05-20 (Estimated); Results first posted 2011-07-14 (Estimated); Last update posted 2021-06-14 (Actual); Status verified 2021-06

CONDITIONS: Major Depressive Disorder
MeSH Terms: conditions — Depressive Disorder, Major | interventions — Antidepressive Agents; Lisdexamfetamine Dimesylate

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Active (Experimental): Antidepressant + SPD489
  Interventions: Drug: Antidepressant + SPD489 (lisdexamfetamine dimesylate)
- Placebo (Placebo Comparator): Antidepressant + placebo
  Interventions: Drug: Antidepressant + placebo

INTERVENTIONS:
Drug: Antidepressant + SPD489 (lisdexamfetamine dimesylate) — Escitalopram oxalate (antidepressant) 20 mg/day oral + 20, 30, or 50 mg SPD489 oral once daily for 6 weeks
  Other Names: LDX, Vyvanse
  Arms: Active
Drug: Antidepressant + placebo — Escitalopram oxalate (antidepressant) 20 mg/day oral + placebo oral once daily for 6 weeks
  Arms: Placebo

SUMMARY:
To evaluate the efficacy of SPD489 when used as augmentation to an antidepressant in the treatment of major depressive disorder (MDD) as measured by mean change in total Montgomery-Ǻsberg Depression Rating Scale (MADRS) scores.

ELIGIBILITY:
Inclusion Criteria:

* Adults aged 18-55 with a primary diagnosis of nonpsychotic MDD

Exclusion Criteria:

* History of non-response to multiple antidepressants

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 246 (Actual)
Dates: Start 2009-07-30 (Actual); Primary Completion 2010-08-04 (Actual); Study Completion 2010-08-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Study Director, Study Director — Takeda
Locations (15):
- United States (15):
  - Pharmacology Research Institute (PRI), Newport Beach, California
  - Affiliated Research Institute, San Diego, California
  - Florida Clinical Research Center, LLC, Bradenton, Florida
  - Gulfcoast Clinical Research Center, Fort Myers, Florida
  - Clinical Neuroscience Solutions, Inc., Orlando, Florida
  - Atlanta Institute of Medicine & Research, Atlanta, Georgia
  - Carman Research, Smyrna, Georgia
  - Vince & Associates Clinical Research, Overland Park, Kansas
  - Duke University Medical Center, Durham, North Carolina
  - North Star Medical Research, LLC, Middleburg Heights, Ohio
  - IPS Research Company, Oklahoma City, Oklahoma
  - Summit Research Network, Portland, Oregon
  - FutureSearch Clinical Trials, LP, Austin, Texas
  - Northwest Clinical Research Center, Bellevue, Washington
  - Summit Research Network (Seattle), LLC, Seattle, Washington

REFERENCES:
- [Result] Trivedi MH, Cutler AJ, Richards C, Lasser R, Geibel BB, Gao J, Sambunaris A, Patkar AA. A randomized controlled trial of the efficacy and safety of lisdexamfetamine dimesylate as augmentation therapy in adults with residual symptoms of major depressive disorder after treatment with escitalopram. J Clin Psychiatry. 2013 Aug;74(8):802-9. doi: 10.4088/JCP.13m08360. PMID 24021497
- See also: FDA Recall Information — http://www.fda.gov/opacom/7alerts.html

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: 246 subjects entered the antidepressant lead-in phase receiving escitalopram oxalate (antidepressant) 20 mg/day for 8 weeks. After 8 weeks, subjects with residual depressive symptoms (n = 177) were randomly assigned (stratified by remission, either remitters or non-remitters) to receive augmentation therapy (either SPD489 or placebo).
Groups:
- Antidepressant + SPD489: Subjects with residual depressive symptoms (symptoms of depression that remain after initial antidepressant treatment) after the 8-week lead-in period with antidepressant (escitalopram @ 20 mg/day) were randomly assigned to receive augmentation therapy (antidepressant @ 20 mg/day + SPD489 @ either 20, 30, or 50 mg/day) for 6 weeks. This includes both non-remitters (Montgomery-Ǻsberg Depression Rating Scale [MADRS] total score greater than 10 at augmentation baseline) and remitters (MADRS total score of less than or equal to 10 at augmentation baseline).
- Antidepressant + Placebo .: Subjects with residual depressive symptoms after the 8-week lead-in period with antidepressant were randomly assigned to receive augmentation therapy (antidepressant @ 20 mg/day + placebo) for 6 weeks. This includes both non-remitters and remitters.
Period: Overall Study
Arm/Group | Antidepressant + SPD489 | Antidepressant + Placebo .
Started | 89 | 88
Completed | 78 | 79
Not Completed | 11 | 9
Not completed — Lost to Follow-up | 3 | 3
Not completed — Withdrawal by Subject | 1 | 2
Not completed — Adverse Event | 4 | 2
Not completed — Non-compliance with study medication | 2 | 0
Not completed — Sponsor decision | 1 | 0
Not completed — Positive urine drug screen | 0 | 1
Not completed — Non-adherence to visit schedule | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Antidepressant + SPD489 | Antidepressant + Placebo . | Total
Number analyzed (Participants) | 88 | 85 | 173
Age, Continuous [Mean (Standard Deviation); unit: years] — 177 subjects were randomized. However, 4 withdrew before receiving any randomized augmentation treatment. Therefore, 173 subjects were included in the Randomized Safety Analysis Set defined as all subjects who took at least 1 dose of randomized augmentation treatment and at least 1 follow-up safety assessment.
  years | 39.4 (9.65) | 38.6 (10.38) | 39.0 (9.99)
Age, Customized [Count of Participants; unit: Participants] — 177 subjects were randomized. However, 4 withdrew before receiving any randomized augmentation treatment. Therefore, 173 subjects were included in the Randomized Safety Analysis Set defined as all subjects who took at least 1 dose of randomized augmentation treatment and at least 1 follow-up safety assessment.
  Participants
    18-40 years | 44 | 49 | 93
    41-55 years | 44 | 36 | 80
Sex: Female, Male [Count of Participants; unit: Participants] — 177 subjects were randomized. However, 4 withdrew before receiving any randomized augmentation treatment. Therefore, 173 subjects were included in the Randomized Safety Analysis Set defined as all subjects who took at least 1 dose of randomized augmentation treatment and at least 1 follow-up safety assessment.
  Participants
    Female | 53 | 54 | 107
    Male | 35 | 31 | 66
Region of Enrollment [Count of Participants; unit: Participants] — 177 subjects were randomized. However, 4 withdrew before receiving any randomized augmentation treatment. Therefore, 173 subjects were included in the Randomized Safety Analysis Set defined as all subjects who took at least 1 dose of randomized augmentation treatment and at least 1 follow-up safety assessment.
  Participants
    United States | 88 | 85 | 173

OUTCOME MEASURES:

1. Primary Outcome: Change From Augmentation Baseline for Non-Remitters in Montgomery-Ǻsberg Depression Rating Scale (MADRS) Total Score at Week 6 - Last Observation Carried Forward (LOCF)
Description: MADRS is a validated, 10-item rating scale with each item being scored on a scale from 0-6 with a total score ranging from 0-60. Lower scores indicate a decreased severity of depression.
Time Frame: Augmentation Baseline, 6 weeks
Population: Primary Efficacy Analysis Set defined as all non-remitters (MADRS total score greater than 10 at augmentation baseline) who take at least 1 dose of randomized augmentation treatment and have at least 1 primary efficacy measurement after randomization.
Measure: Least Squares Mean (Standard Error); unit: Units on a scale
Groups:
- Antidepressant + SPD489 (Non-remitters): Subjects with residual depressive symptoms after the 8-week lead-in period with antidepressant were randomly assigned to receive augmentation therapy (SPD489). At augmentation baseline, randomization was stratified by Non-remitters and remitters. Non-remitters were defined as subjects who had an MADRS total score of greater than 10 at augmentation baseline. Subjects received antidepressant (escitalopram @ 20 mg/day) + an optimal dose of SPD489 (either 20, 30, or 50 mg/day) for 6 weeks.
- Antidepressant + Placebo (Non-remitters): Subjects with residual depressive symptoms after the 8-week lead-in period with antidepressant were randomly assigned to receive augmentation therapy (placebo). At augmentation baseline, randomization was stratified by Non-remitters and remitters. Non-remitters were defined as subjects who had an MADRS total score of greater than 10 at augmentation baseline. Subjects received antidepressant (escitalopram @ 20 mg/day) + placebo for 6 weeks.
Arm/Group | Antidepressant + SPD489 (Non-remitters) | Antidepressant + Placebo (Non-remitters)
Number analyzed (Participants) | 65 | 64
Units on a scale | -7.1 (0.93) | -4.9 (0.94)
Statistical Analysis 1: Comparison: Antidepressant + SPD489 (Non-remitters) vs Antidepressant + Placebo (Non-remitters); Test type: Superiority or Other; p = 0.0902, ANCOVA — The test was performed a priori at the significance level of 0.10; Mean Difference (Final Values) = -2.3, 90% CI 2-sided [-4.5 to -0.1]

2. Secondary Outcome: Change From Augmentation Baseline for Non-Remitters in the Hamilton Depression Scale (HAM-D) Total Score at Week 6 - LOCF
Description: The HAM-D is a validated rating scale which consists of 17 items. Nine of the items are scored on a scale of 0-4 and 8 items are scored on a scale of 0-2 for a total scoring range of 0-52. A score of 0-7 is generally accepted to be within the normal range (or in clinical remission), while a score of 20 or higher indicates increased severity of depression. In general, the lower the total score the less severe the depression.
Time Frame: Augmentation Baseline, 6 weeks
Population: Primary Efficacy Analysis Set
Measure: Least Squares Mean (Standard Error); unit: Units on a scale
Arm/Group | Antidepressant + SPD489 (Non-remitters) | Antidepressant + Placebo (Non-remitters)
Number analyzed (Participants) | 65 | 64
Units on a scale | -4.9 (0.64) | -4.0 (0.65)
Statistical Analysis 1: Comparison: Antidepressant + SPD489 (Non-remitters) vs Antidepressant + Placebo (Non-remitters); Test type: Superiority or Other; p = 0.3091, ANCOVA — The test was performed a priori at the significance level of 0.10; Mean Difference (Final Values) = -0.9, 90% CI 2-sided [-2.4 to 0.6]

3. Secondary Outcome: Change From Augmentation Baseline for Non-Remitters in the Sheehan Disability Scale (SDS) Total Score at Week 6
Description: Designed to evaluate the extent to which illness symptoms impact a subject's life in 3 areas: work/school, social, and family/home. Each area is scored on a scale from 0 (no impairment) to 10 (highly impaired) with a total score ranging from 0 (unimpaired) to 30 (highly impaired). Lower scores translate into less impairment.
Time Frame: Augmentation Baseline, 6 weeks
Population: Primary Efficacy Analysis Set
Measure: Least Squares Mean (Standard Error); unit: Units on a scale
Arm/Group | Antidepressant + SPD489 (Non-remitters) | Antidepressant + Placebo (Non-remitters)
Number analyzed (Participants) | 63 | 62
Units on a scale | -3.7 (0.73) | -1.7 (0.74)
Statistical Analysis 1: Comparison: Antidepressant + SPD489 (Non-remitters) vs Antidepressant + Placebo (Non-remitters); Test type: Superiority or Other; p = 0.0573, ANCOVA — The test was performed a priori at the significance level of 0.10; Mean Difference (Final Values) = -2.0, 90% CI 2-sided [-3.7 to -0.3]

4. Secondary Outcome: Percentage of Non-Remitters With Improvement on Clinical Global Impression-Improvement (CGI-I) at Week 6 - LOCF
Description: Clinical Global Impression-Improvement (CGI-I) consists of a 7-point scale ranging from 1 (very much improved) to 7 (very much worse). Improvement is defined as a score of 1 (very much improved) or 2 (much improved) on the scale.
Time Frame: 6 weeks
Population: Primary Efficacy Analysis Set
Measure: Number; unit: Percent of Participants
Arm/Group | Antidepressant + SPD489 (Non-remitters) | Antidepressant + Placebo (Non-remitters)
Number analyzed (Participants) | 65 | 64
Percent of Participants | 60.0 | 45.3
Statistical Analysis 1: Comparison: Antidepressant + SPD489 (Non-remitters) vs Antidepressant + Placebo (Non-remitters); Test type: Superiority or Other; p = 0.2368, Cochran-Mantel-Haenszel

5. Secondary Outcome: Assessment in Non-Remitters of Clinical Global Impression-Severity of Illness (CGI-S) at Augmentation Baseline
Description: CGI-S assesses the severity of the subject's condition on a 7-point scale ranging from 1 (normal, not at all ill) to 7 (among the most extremely ill)
Time Frame: Augmentation baseline
Population: Primary Efficacy Analysis Set
Measure: Number; unit: Percent of participants
Arm/Group | Antidepressant + SPD489 (Non-remitters) | Antidepressant + Placebo (Non-remitters)
Number analyzed (Participants) | 64 | 64
Percent of participants
  Normal, not at all ill | 1.5 | 1.6
  Borderline mentally ill | 20.0 | 12.5
  Mildly ill | 40.0 | 34.4
  Moderately ill | 32.3 | 48.4
  Markedly ill | 6.2 | 3.1
  Severely ill | 0 | 0
  Among the most extremely ill | 0 | 0

6. Secondary Outcome: Assessment in Non-Remitters of Clinical Global Impression-Severity of Illness (CGI-S) at Week 6
Description: as for outcome 5
Time Frame: 6 weeks
Population: Primary Efficacy Analysis Set
Measure: Number; unit: Percent of participants
Arm/Group | Antidepressant + SPD489 (Non-remitters) | Antidepressant + Placebo (Non-remitters)
Number analyzed (Participants) | 63 | 62
Percent of participants
  Normal, not at all ill | 27.0 | 14.5
  Borderline mentally ill | 31.7 | 24.2
  Mildly ill | 30.2 | 22.6
  Moderately ill | 9.5 | 29.0
  Markedly ill | 1.6 | 9.7
  Severely ill | 0 | 0
  Among the most extremely ill | 0 | 0

7. Secondary Outcome: Change From Augmentation Baseline for Non-Remitters in the Behavior Rating Inventory of Executive Function - Adult Version (BRIEF-A) Scale Total Score at Week 6
Description: BRIEF-A is a validated 75-item questionnaire composed of three scales (Global Executive Composite, Behavioral Recognition Index, and Metacognition Index). Items are rated 1 (never), 2 (sometimes), and 3 (often). There is no range for a total score. Raw scale scores are used to develop interpretive reports. Lower scores reflect better functioning.
Time Frame: Augmentation Baseline and 6 weeks
Population: Primary Efficacy Analysis Set
Measure: Least Squares Mean (Standard Error); unit: Units on a scale
Arm/Group | Antidepressant + SPD489 (Non-remitters) | Antidepressant + Placebo (Non-remitters)
Number analyzed (Participants) | 62 | 60
Units on a scale
  Global Executive Composite | -4.7 (1.03) | -1.7 (1.04)
  Behavioral Regulation Index | -3.7 (0.97) | -1.7 (0.99)
  Metacognition Index | -4.8 (1.04) | -1.5 (1.06)
Statistical Analysis 1: Comparison: Antidepressant + SPD489 (Non-remitters) vs Antidepressant + Placebo (Non-remitters); Global Executive Composite; Test type: Superiority or Other; p = 0.0463, ANCOVA — The test was performed a priori at the significance level of 0.10; Mean Difference (Final Values) = -3.0, 90% CI 2-sided [-5.4 to -0.5]
Statistical Analysis 2: Comparison: Antidepressant + SPD489 (Non-remitters) vs Antidepressant + Placebo (Non-remitters); Behavioral Regulation Index; Test type: Superiority or Other; p = 0.1431, ANCOVA — The test was performed a priori at the significance level of 0.10; Mean Difference (Final Values) = -2.0, 90% CI 2-sided [-4.3 to 0.3]
Statistical Analysis 3: Comparison: Antidepressant + SPD489 (Non-remitters) vs Antidepressant + Placebo (Non-remitters); Metacognition Index; Test type: Superiority or Other; p = 0.0281, ANCOVA — The test was performed a priori at the significance level of 0.10; Mean Difference (Final Values) = -3.3, 90% CI 2-sided [-5.8 to -0.8]

8. Secondary Outcome: Change From Augmentation Baseline for Non-Remitters in the Multidimensional Assessment of Fatigue (MAF) Scale Total Score at Week 6
Description: MAF contains 16 items scored on a scale from 1 (not at all) to 10 (a great deal). Answers are converted to a Global Fatigue Index with total scores ranging from 1 (no fatigue) to 50 (severe fatigue). Lower scores indicate less fatigue.
Time Frame: Augmentation Baseline and 6 weeks
Population: Primary Efficacy Analysis Set
Measure: Least Squares Mean (Standard Error); unit: Units on a scale
Arm/Group | Antidepressant + SPD489 (Non-remitters) | Antidepressant + Placebo (Non-remitters)
Number analyzed (Participants) | 63 | 62
Units on a scale | -5.3 (1.25) | -2.3 (1.26)
Statistical Analysis 1: Comparison: Antidepressant + SPD489 (Non-remitters) vs Antidepressant + Placebo (Non-remitters); Test type: Superiority or Other; p = 0.0920, ANCOVA — The test was performed a priori at the significance level of 0.10; Mean Difference (Final Values) = -3.0, 90% CI 2-sided [-6.0 to -0.1]

9. Secondary Outcome: Change From Augmentation Baseline for Non-Remitters in the Quick Inventory of Depressive Symptomatology - Self-Report (QIDS-SR) Scale Total Score at Week 6
Description: QIDS-SR is a validated, self-reported rating scale that contains 16 items scored on a scale from 0-3 with total scores ranging from 0 (no depression) to 27 (very severe depression). Lower scores indicate less depression.
Time Frame: Augmentation Baseline and 6 weeks
Population: Primary Efficacy Analysis Set
Measure: Least Squares Mean (Standard Error); unit: Units on a scale
Arm/Group | Antidepressant + SPD489 (Non-remitters) | Antidepressant + Placebo (Non-remitters)
Number analyzed (Participants) | 63 | 62
Units on a scale | -2.4 (0.45) | -1.2 (0.46)
Statistical Analysis 1: Comparison: Antidepressant + SPD489 (Non-remitters) vs Antidepressant + Placebo (Non-remitters); Test type: Superiority or Other; p = 0.0774, ANCOVA — The test was performed a priori at the significance level of 0.10; Mean Difference (Final Values) = -1.2, 90% CI 2-sided [-2.2 to -0.1]

10. Secondary Outcome: Change From Augmentation Baseline for Remitters in MADRS Total Score at Week 6 - LOCF
Description: as for outcome 1
Time Frame: Augmentation Baseline and 6 weeks
Population: Full Analysis Set (FAS) defined as all subjects who take at least 1 dose of randomized augmentation treatment and have at least 1 primary efficacy measurement after randomization.
Measure: Least Squares Mean (Standard Error); unit: Units on a scale
Groups:
- Antidepressant + SPD489 (Remitters): Subjects with residual depressive symptoms after the 8-week lead-in period with antidepressant were randomly assigned to receive augmentation therapy (SPD489). At augmentation baseline, randomization was stratified by non-remitters and remitters. Remitters were defined as subjects who had an MADRS total score of less than or equal to 10 at augmentation baseline. Subjects received antidepressant (escitalopram @ 20 mg/day) + an optimal dose of SPD489 (either 20, 30, or 50 mg/day) for 6 weeks.
- Antidepressant + Placebo (Remitters): Subjects with residual depressive symptoms after the 8-week lead-in period with antidepressant were randomly assigned to receive augmentation therapy (placebo). At augmentation baseline, randomization was stratified by non-remitters and remitters. Remitters were defined as subjects who had an MADRS total score of less than or equal to 10 at augmentation baseline. Subjects received antidepressant (escitalopram @ 20 mg/day) + placebo for 6 weeks.
Arm/Group | Antidepressant + SPD489 (Remitters) | Antidepressant + Placebo (Remitters)
Number analyzed (Participants) | 23 | 21
Units on a scale | 0.1 (1.13) | -1.1 (1.18)
Statistical Analysis 1: Comparison: Antidepressant + SPD489 (Remitters) vs Antidepressant + Placebo (Remitters); Test type: Superiority or Other; p = 0.4726, ANCOVA — The test was performed a priori at the significance level of 0.10; Mean Difference (Final Values) = 1.2, 90% CI 2-sided [-1.6 to 4.0]

11. Secondary Outcome: Change From Augmentation Baseline for Remitters in the HAM-D Total Score at Week 6 - LOCF
Description: as for outcome 2
Time Frame: Augmentation Baseline and 6 weeks
Population: FAS
Measure: Least Squares Mean (Standard Error); unit: Units on a scale
Arm/Group | Antidepressant + SPD489 (Remitters) | Antidepressant + Placebo (Remitters)
Number analyzed (Participants) | 23 | 21
Units on a scale | -0.8 (0.92) | -1.6 (0.96)
Statistical Analysis 1: Comparison: Antidepressant + SPD489 (Remitters) vs Antidepressant + Placebo (Remitters); Test type: Superiority or Other; p = 0.5182, ANCOVA — The test was performed a priori at the significance level of 0.10; Mean Difference (Final Values) = 0.9, 90% CI 2-sided [-1.4 to 3.1]

12. Secondary Outcome: Change From Augmentation Baseline for Remitters in the SDS Total Score at Week 6
Description: as for outcome 3
Time Frame: Augmentation Baseline and 6 weeks
Population: FAS
Measure: Least Squares Mean (Standard Error); unit: Units on a scale
Arm/Group | Antidepressant + SPD489 (Remitters) | Antidepressant + Placebo (Remitters)
Number analyzed (Participants) | 22 | 21
Units on a scale | -1.6 (0.89) | -0.6 (0.91)
Statistical Analysis 1: Comparison: Antidepressant + SPD489 (Remitters) vs Antidepressant + Placebo (Remitters); Test type: Superiority or Other; p = 0.4630, ANCOVA — The test was performed a priori at the significance level of 0.10; Mean Difference (Final Values) = -0.9, 90% CI 2-sided [-3.1 to 1.2]

13. Secondary Outcome: Percentage of Remitters With Improvement on CGI-I at Week 6 - LOCF
Description: as for outcome 4
Time Frame: 6 weeks
Population: FAS
Measure: Number; unit: Percent of participants
Arm/Group | Antidepressant + SPD489 (Remitters) | Antidepressant + Placebo (Remitters)
Number analyzed (Participants) | 23 | 21
Percent of participants | 65.2 | 52.4
Statistical Analysis 1: Comparison: Antidepressant + SPD489 (Remitters) vs Antidepressant + Placebo (Remitters); Test type: Superiority or Other; p = 0.5230, Cochran-Mantel-Haenszel

14. Secondary Outcome: Assessment in Remitters of CGI-S at Augmentation Baseline
Description: as for outcome 5
Time Frame: Augmentation Baseline
Population: FAS
Measure: Number; unit: Percent of participants
Arm/Group | Antidepressant + SPD489 (Remitters) | Antidepressant + Placebo (Remitters)
Number analyzed (Participants) | 23 | 21
Percent of participants
  Normal, not at all ill | 26.1 | 23.8
  Borderline mentally ill | 47.8 | 71.4
  Mildly ill | 21.7 | 4.8
  Moderately ill | 4.3 | 0
  Markedly ill | 0 | 0
  Severely ill | 0 | 0
  Among the most extremely ill | 0 | 0

15. Secondary Outcome: Assessment in Remitters of CGI-S at Week 6
Description: as for outcome 5
Time Frame: 6 weeks
Population: FAS
Measure: Number; unit: Percent of participants
Arm/Group | Antidepressant + SPD489 (Remitters) | Antidepressant + Placebo (Remitters)
Number analyzed (Participants) | 22 | 21
Percent of participants
  Normal, not at all ill | 50.0 | 61.9
  Borderline mentally ill | 36.4 | 23.8
  Mildly ill | 13.6 | 9.5
  Moderately ill | 0 | 4.8
  Markedly ill | 0 | 0
  Severely ill | 0 | 0
  Among the most extremely ill | 0 | 0

16. Secondary Outcome: Change From Augmentation Baseline for Remitters in the BRIEF-A Scale Total Score at Week 6
Description: BRIEF-A is a validated 86-item questionnaire composed of three scales (Global Executive Composite, Behavioral Recognition Index, and Metacognition Index). Items are rated 1 (never), 2 (sometimes), and 3 (often). Lower scores reflect better functioning.
Time Frame: Augmentation baseline and 6 weeks
Population: FAS
Measure: Least Squares Mean (Standard Error); unit: Units on a scale
Arm/Group | Antidepressant + SPD489 (Remitters) | Antidepressant + Placebo (Remitters)
Number analyzed (Participants) | 21 | 21
Units on a scale
  Global Executive Composite | -0.9 (1.21) | -2.7 (1.21)
  Behavioral Regulation Index | -0.4 (1.37) | -1.5 (1.37)
  Metacognition Index | -1.1 (1.24) | -3.4 (1.24)
Statistical Analysis 1: Comparison: Antidepressant + SPD489 (Remitters) vs Antidepressant + Placebo (Remitters); Global Executive Composite; Test type: Superiority or Other; p = 0.2876, ANCOVA — The test was performed a priori at the significance level of 0.10; Mean Difference (Final Values) = 1.8, 90% CI 2-sided [-1.0 to 4.7]
Statistical Analysis 2: Comparison: Antidepressant + SPD489 (Remitters) vs Antidepressant + Placebo (Remitters); Behavioral Regulation Index; Test type: Superiority or Other; p = 0.5590, ANCOVA — The test was performed a priori at the significance level of 0.10; Mean Difference (Final Values) = 1.1, 90% CI 2-sided [-2.1 to 4.4]
Statistical Analysis 3: Comparison: Antidepressant + SPD489 (Remitters) vs Antidepressant + Placebo (Remitters); Metacognition Index; Test type: Superiority or Other; p = 0.2079, ANCOVA — The test was performed a priori at the significance level of 0.10; Mean Difference (Final Values) = 2.3, 90% CI 2-sided [-0.7 to 5.2]

17. Secondary Outcome: Change From Augmentation Baseline for Remitters in the MAF Scale Total Score at Week 6
Description: as for outcome 8
Time Frame: Augmentation baseline and 6 weeks
Population: FAS
Measure: Least Squares Mean (Standard Error); unit: Units on a scale
Arm/Group | Antidepressant + SPD489 (Remitters) | Antidepressant + Placebo (Remitters)
Number analyzed (Participants) | 22 | 21
Units on a scale | -4.0 (1.77) | -0.2 (1.81)
Statistical Analysis 1: Comparison: Antidepressant + SPD489 (Remitters) vs Antidepressant + Placebo (Remitters); Test type: Superiority or Other; p = 0.1489, ANCOVA — The test was performed a priori at the significance level of 0.10; Mean Difference (Final Values) = -3.7, 90% CI 2-sided [-8.0 to 0.5]

18. Secondary Outcome: Change From Augmentation Baseline for Remitters in the QIDS-SR Scale Total Score at Week 6
Description: as for outcome 9
Time Frame: Augmentation baseline and 6 weeks
Population: FAS
Measure: Least Squares Mean (Standard Error); unit: Units on a scale
Arm/Group | Antidepressant + SPD489 (Remitters) | Antidepressant + Placebo (Remitters)
Number analyzed (Participants) | 22 | 21
Units on a scale | -1.9 (0.57) | -0.4 (0.58)
Statistical Analysis 1: Comparison: Antidepressant + SPD489 (Remitters) vs Antidepressant + Placebo (Remitters); Test type: Superiority or Other; p = 0.0852, ANCOVA — The test was performed a priori at the significance level of 0.10; Mean Difference (Final Values) = -1.4, 90% CI 2-sided [-2.8 to -0.1]

ADVERSE EVENTS:
Description: Randomized Safety Analysis Set (RSAS) defined as all subjects who take at least 1 dose of randomized augmentation treatment and at least 1 follow-up safety assessment.
Arm/Group | Antidepressant + SPD489 | Antidepressant + Placebo .
Serious Adverse Events (participants affected / at risk) | 0/88 | 1/85
Other Adverse Events (participants affected / at risk) | 35/88 | 15/85
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Antidepressant + SPD489 (N=88) | Antidepressant + Placebo . (N=85)
Rhabdomyolysis (Musculoskeletal and connective tissue disorders) | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Antidepressant + SPD489 (N=88) | Antidepressant + Placebo . (N=85)
Dry mouth (Gastrointestinal disorders) | 10 | 0
Headache (Nervous system disorders) | 10 | 4
Decreased appetite (Metabolism and nutrition disorders) | 6 | 2
Nasopharyngitis (Infections and infestations) | 5 | 3
Insomnia (Psychiatric disorders) | 4 | 6

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
If a multicenter publication is not submitted within twelve (12) months after conclusion, abandonment or termination of the Study at all sites, or after Sponsor confirms there shall be no multicenter Study publication, the Institution and/or such Principal Investigator may publish the results from the Institution site individually.